CLINICAL TRIAL: NCT02310204
Title: Evaluation of a Therapeutic Education Program in Patients With Moderate to Severe Psoriasis : a Multicenter Randomized Controlled Study
Brief Title: Therapeutic Education Program in Psoriasis
Acronym: EDUPSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10 141 01
Record Dates: First submitted 2014-12-01; First posted 2014-12-08 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- multidisciplinary education program (Experimental): individual and group education sessions over a 6-month period
  Interventions: Behavioral: multidisciplinary education program
- Standard psoriasis care alone (Active Comparator): Standard psoriasis care alone
  Interventions: Other: standard psoriasis care alone

INTERVENTIONS:
Behavioral: multidisciplinary education program — both individual and group education sessions over a 6-month period in addition to standard psoriasis care
  Arms: multidisciplinary education program
Other: standard psoriasis care alone
  Arms: Standard psoriasis care alone

SUMMARY:
The primary objective of this research protocol is to assess the effect of a structured therapeutic education program on the quality of life of patients with moderate to severe psoriasis

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory skin disease affecting 1 to 3% of the French population. Moderate to severe psoriasis has a significant impact on quality of life. Psoriasis is associated with an increased risk of depression, social isolation, unemployment. In addition, it has recently be shown that patients with moderate to severe psoriasis have an increased incidence of cardiovascular risk factors such as hypertension, overweight, hyperlipidemia and exposure to tobacco and alcohol. These so-called comorbidites may have a negative impact on psoriasis management. They also may account for the reduced life expectancy reported in patients with severe psoriasis. Therapeutic education is a structured process whose objective is to help patients to acquire or to maintain competencies that are required to live with a chronic disease. Therapeutic education is an important process to be integrated into the therapeutic strategy. It has to take into account co-morbidities, social and psychological context and its priorities need to be defined with the patient.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe psoriasis defined as patients receiving a systemic psoriasis treatment including methotrexate, cyclosporine, PUVA, retinoids or a biological agent and with significant impact on quality of life defined as a Skindex > 18
* Patients with palmo-plantar or erythrodermic psoriasis may be included if they can be classified as moderate to severe according the above described definitions

Exclusion Criteria:

* Patients not able to give informed consent,
* Patients not able to follow the program,
* Patients without social security affiliation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
skindex quality of life | 3 months
  evaluation of quality of life

SECONDARY OUTCOMES:
SF36 - Short Form 36 | 3 MONTHS
PASI - Psoriasis Area and Severity Index | 3 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Carle PAUL, MD, Principal Investigator — University Hospital, Toulouse
Locations (9):
- France (9):
  - University Hospital, Brest
  - Edouard Herriot, Lyon
  - Unversity Hospital, Lyon
  - Timone Hospital, Marseille
  - Saint Joseph Hospital, Marseille
  - University Hospital, Nantes
  - Archet Hospital, Nice
  - Saint-Louis Hospital, Paris
  - Haut Leveque Hospital, Pessac

REFERENCES:
- [Background] Viguier M, Livideanu C, Beylot-Barry M, Richard MA, Paul C, Bachelez H, Aubin F; Groupe de Recherche sur le Psoriasis. Observational case series on a group of psoriasis patients who failed to respond to any TNF blockers. J Dermatolog Treat. 2014 Feb;25(1):75-7. doi: 10.3109/09546634.2013.806766. Epub 2013 Jun 20. PMID 23724854
- [Result] Jendoubi F, Balica S, Richard MA, Chiaverini C, Bernier C, Quiles N, Bachelez H, Beylot-Barry M, Mallet S, Goujon C, Parier J, Misery L, Carrere F, Lauwers-Cances V, Paul C; French Psoriasis Research Group. A Multicentre Randomised Controlled Study Evaluating the Effect of a Standardised Education Programme on Quality of Life, Disease Severity, and Disease Knowledge in Patients with Moderate-To-Severe Psoriasis: The EDUPSO Study. Dermatology. 2022;238(4):630-639. doi: 10.1159/000520289. Epub 2021 Dec 9. PMID 34883480